CLINICAL TRIAL: NCT02472418
Title: A Multi-Center, Randomized, Placebo-Controlled, Double-Blind, Crossover Study Evaluating Efficacy of DFN-15 in Patients With Migraine Headache With or Without Aura
Brief Title: Two Dose Levels of DFN-15 vs. Placebo in Patients With Migraine Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DFN-15-CD-002
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- DFN-15 120 mg (treatment A) (Experimental): DFN-15 120 mg (treatment A)
  Interventions: Drug: DFN-15 Dose A (treatment A)
- DFN-15 240 mg (treatment B) (Experimental): DFN-15 240 mg (treatment B)
  Interventions: Drug: DFN-15 Dose B (treatment B)
- Placebo (treatment C) (Placebo Comparator): Placebo (treatment C)
  Interventions: Other: Placebo (treatment C)

INTERVENTIONS:
Drug: DFN-15 Dose A (treatment A) — DFN-15 Dose A administered
  Other Names: DFN-15 120 mg
  Arms: DFN-15 120 mg (treatment A)
Drug: DFN-15 Dose B (treatment B) — DFN-15 Dose B administered
  Other Names: DFN-15 240 mg
  Arms: DFN-15 240 mg (treatment B)
Other: Placebo (treatment C) — Placebo administered
  Other Names: Placebo (no active ingredient)
  Arms: Placebo (treatment C)

SUMMARY:
Crossover study of DFN-15 dose A versus DFN-15 dose B versus Placebo in the treatment of migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of episodic migraine (as defined by International Classification of Headache Disorders [ICHD]-228) who experience an average of 2 to 6 migraine attacks a month for the past 12 months with no more than 14 headache days per month, and with at least 48 hours of headache-free time between migraine attacks;
2. Patients with onset of migraine with or without aura before age 50;
3. Patients who have migraine with or without aura, in which the aura cannot last longer than 60 minutes;
4. Patients who report usual migraine pain of 2 (moderate) or 3 (severe) on headache pain severity scale.

Exclusion Criteria:

1. Patients with medication overuse headache (MOH) as defined by ICHD-228:

   * Opioids ≥ 10 days a month during the 90 days prior to screening
   * Combination medications (eg, Fiorinal® ≥ 10 days a month)
   * Nonsteroidal anti-inflammatory drugs (NSAIDs) or other simple medications > 14 days a month during the 90 days prior to screening
   * Triptans or ergots ≥ 10 days a month during the 90 days prior to screening
2. Patients on chronic warfarin sodium;
3. Patients taking monoamine oxidase-A (MAO-A) inhibitors;
4. Patients on unstable dosages of chronic medications during the 3 months prior to and through screening, or who are not willing or able to maintain a stable pre-study dose throughout study participation;
5. Patients with more than 6 migraine attacks a month and/or more than 14 headache days a month (based upon patient self-report);
6. Patients with hemiplegic migraine or migraine with brain stem aura or other forms of neurologically complicated migraine;
7. Patients with atypical aura;
8. Patients with prolonged aura (more than 1 hour).
9. Patients with a history of stroke or transient ischemic attack;
10. Patients with a history of migralepsy or a concurrent diagnosis of seizure disorder;
11. Patients who cannot differentiate between a migraine headache and a tension-type or cluster headache or any other non-migraine headache;
12. Patients with a history of more than 10 tension-type headaches per month;
13. Patients with a history of cluster headache;
14. Patients with a diagnosis of ICHD-2 "probable migraine";
15. Patients with uncontrolled hypertension (screening blood pressure ≥ 140/90 mmHg despite appropriate pharmacotherapy);
16. Patients with severe renal impairment (defined as serum creatinine > 1.9 mg/dL);
17. Patients with serum total bilirubin > 1.9 mg/dL;
18. Patients with serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 3 times the upper limit of normal;
19. Patients with positive serology for human immunodeficiency virus (HIV), Hepatitis B surface antigen, Hepatitis C antibody.
20. Patients with a history of alcohol or substance abuse (including marijuana and medical marijuana) within 1 year that would compromise data collection;
21. Patients with a history of or current neurological or psychiatric impairment, or cognitive dysfunction that, in the opinion of the investigator, would compromise data collection;
22. Patients with any other medical condition that, in the judgment of the investigator or medical monitor, would confound the objectives of the study (eg, cancer history [except basal cell carcinoma], systemic lupus erythematosus);
23. Patients who have participated in a clinical trial involving any medication during the past 30 days or 5 half-lives of the study medication, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Pain Free, defined as a score of "0" on a numerical scale of "0" to "3" | 2 hour
  Percentage of subjects who are migraine headache free at 2 hours after taking study drug administration

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - California Medical Clinic for Headache, Santa Monica, California
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinvest/ A Division of Banyan Group, Inc., Springfield, Missouri
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico

REFERENCES:
- [Result] Munjal S, Bennett A. Efficacy and safety of DFN-15, an oral liquid formulation of celecoxib, in adults with migraine: a multicenter, randomized, placebo-controlled, double-blind, crossover study. Neuropsychiatr Dis Treat. 2017 Nov 7;13:2797-2802. doi: 10.2147/NDT.S151834. eCollection 2017. PMID 29158678